CLINICAL TRIAL: NCT03731403
Title: Remineralization Potential of MI Varnish(CPP-ACP and Fluoride) Versus Fluoride Varnish in Controlling White Spot Lesions in Maxillary Primary Incisors: A Randomized Clinical Trial
Brief Title: Remineralization Potential of MI Varnish Versus Fluoride Varnish on White Spot Lesions in Maxillary Primary Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Sayed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-28-10-2017
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Remineralization Effect of the Varnish on White Spot Lesions
Keywords: Early childhood caries; Casein phosphopeptides-amorphous calcium phosphate; fluoride; remineralization potential; varnish
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Fluorides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI Varnish (Experimental)
  Interventions: Other: MI varnish
- Profluorid Varnish (Active Comparator)
  Interventions: Other: MI varnish

INTERVENTIONS:
Other: MI varnish — CPP- ACP with 5 % sodium fluoride GC
  Other Names: CPP- ACP with fluoride

SUMMARY:
Remineralization effect of CPP-ACP and Fluoride (MI varnish) versus Fluoride varnish on white spot lesions in maxillary primary incisors

DETAILED DESCRIPTION:
Early childhood caries (ECC) is a very common and consequential chronic disease affecting young children ( Çolak et al., 2013). The prevalence of ECC in Egypt is high, it is about (78%) according to the last Egyptian Report, 2014.

ECC begins with white-spot lesions, and caries can progress continuously, leading to complete destruction of the crown. Calcium and phosphate ions are more readily lost for children because lower mineralization of deciduous enamel. The disease usually develops very quickly and causes many childhood health problems, such as caries-related toothache and infection.

Demineralization and remineralization are dynamic processes in caries initiation, progression, and reversal. Therefore, regulation of the demineralization- remineralization balance is a key to caries prevention and treatment. The ideal method of increasing remineralization is reconstructing the depleted tissues with hydroxyapatite, which is the same inorganic component as the enamel.

Fluoride varnishes have been the standard practice for the professional application of fluoride.

Casien PhosphoPeptide (CPP) is a sticky protein that binds and stabilizes calcium and phosphate ions in an amorphous state. CPP-ACP has been shown to adhere to teeth surfaces.

ELIGIBILITY:
Inclusion Criteria:

1. Children with white spot lesions on their incisors.
2. Age ranging 3-5 years.
3. Good general health.

Exclusion Criteria:

1. Chronic use of medications or antibiotics 2. lack of cooperation in the oral examination 3. Allergies to milk protein or benzoate preservatives 4. Presence of oral soft-tissue lesions or enamel hypoplasia at baseline examination, 5. Children who have received a fluoride supplement or professional topical fluoride application at least 3 months before or during the study period.

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Caries activity | Change from base line, after application at 3, 6, 9 last follow up 12 months
  Measured by ICDAS II

SECONDARY OUTCOMES:
Remineralization | Change from base line, after application at 3, 6, 9 last follow up 12 months
  Measured by EDI

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No